CLINICAL TRIAL: NCT00448786
Title: An Open-Label, Randomized, Phase 1b Study Evaluating the Effect of Different Doses of AMG 706 on the Gallbladder in Subjects With Advanced Solid Tumors
Brief Title: Effect of Different Doses of AMG 706 on the Gallbladder in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20060443
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Solid Tumors
Keywords: gallbladder; AMG 706; solid tumors; Phase 1b; Amgen
MeSH Terms: interventions — motesanib diphosphate

ARMS (3):
- Arm C (Other): Arm C - AMG 706 75 mg BID 5-days on and 2-days off
  Interventions: Drug: AMG 706
- Arm B (Other): Arm B - AMG 706 75 mg BID 2-weeks on and 1-week off
  Interventions: Drug: AMG 706
- Arm A (Other): Arm A = AMG 706 125 mg PO daily continuously
  Interventions: Drug: AMG 706

INTERVENTIONS:
Drug: AMG 706 — Arm B - AMG 706 75 mg BID 2-weeks on and 1-week off
  Arms: Arm B
Drug: AMG 706 — Arm C - 75 mg BID 5-days on, 2-days off
  Arms: Arm C
Drug: AMG 706 — AMG 706 125 mg daily continuously (Arm A)
  Arms: Arm A

SUMMARY:
The study involves the use of three different dosing regimens of AMG 706 in patients with advanced solid tumors to see how the drug affects the gallbladder size and function. The study will be conducted in 11 sites in the US and Australia. A total of 48 patients will be enrolled in the study with the possibility of enrolling 8 more in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced metastatic solid tumor
* Ineligible to receive or progressed on standard of care therapies
* Measurable or non-measurable disease per modified RECIST
* Gallbladder must be in situ on screening ultrasound
* ECOG Performance Status of 0 to 2
* Life expectancy of 6 months or more as determined by the investigator
* Adequate organ and hematologic function as evidenced by laboratory studies prior to randomization
* Men and women 18 years or older

Exclusion Criteria:

* Uncontrolled CNS metastases
* Known history of prior cholecystitis, prior biliary procedure or prior or ongoing biliary disease
* Radiation therapy within 14 days prior to randomization
* Peripheral neuropathy > Grade 1 per CTC AE v.3
* Currently or previously treated with AMG 706 or other VEGF inhibitors such as SU11248 (sunitinib), PTK787 (vatalanib), AZD2171, BAY 43-9006 (sorafenib), ZD6474 (vandetanib)
* Previous treatment with bevacizumab is allowed if at least 6 weeks have elapsed from the last dose of bevacizumab to the date of randomization
* Any anti-coagulant therapy within 7 days prior to randomization; low dose heparin and warfarin for prophylaxis against central venous catheter thrombosis is allowed
* Less than 30 days have elapsed since participation in an investigational drug/device study or currently receiving investigational treatments
* History of arterial or venous thrombosis within 1 year prior to randomization
* History of bleeding diathesis or bleeding within 14 days of randomization
* MI, CVA, TIA, PTCA/stent, CHF, Grade 2 or greater PVD, uncontrolled arrhythmias or unstable angina within one year prior to randomization
* Uncontrolled HTN defined by a resting BP of >150/90 mmHg
* Surgery: major surgical procedure within 4 weeks or 28 days prior to randomization; minor surgical procedure, placement of access device or fine needle aspiration within 7 days of randomization; planned elective surgery while on study
* Non-healing or open wound, ulcer or fracture
* Known ongoing or active infection
* Known (+) for HIV, Hep C or Hep B surface antigen
* Known chronic hepatitis
* Known history of allergy or hypersensitivity to AMG 706 or any of its components
* Pregnant, ie, (+) b-HCG; breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Average change from baseline in gallbladder size (volume by ultrasound) | Anticipated 8 months of treatment with AMG 706
Average change from baseline in gallbladder function (ejection fraction) | Subject treatment with AMG 706 anticipated to be 8 months

SECONDARY OUTCOMES:
Average changes from baseline in gallbladder size (volume by CT scan) | Subject treatment with AMG 706 anticipated to be 8 months
Maximum change from baseline in gallbladder size (volume) and function (ejection fraction) | Subject treatment with AMG 706 anticipated to be 8 months
Change in gallbladder size (volume) and function (ejection fraction) between the last on-treatment measurement and the last available off-treatment measurement | Subject treatment with AMG 706 anticipated to be 8 months
Objective response in subjects with measurable disease at baseline | Subject treatment with AMG 706 anticipated to be 8 months
Pharmacokinetics of AMG 706 monotherapy | Subject treatment with AMG 706 anticipated to be 8 months
Subject incidence of treatment-emergent adverse events (including all, serious, grade 3, grade 4 and treatment-related | Subject treatment with AMG 706 anticipated to be 8 months
Other selected gallbladder characteristics such as size, area, wall thickness, ductal size, presence of stones, pericholecystic fluid and sludge | Subject treatment with AMG 706 anticipated to be 8 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Rosen LS, Lipton L, Price TJ, Belman ND, Boccia RV, Hurwitz HI, Stephenson JJ Jr, Wirth LJ, McCoy S, Hei YJ, Hsu CP, Tebbutt NC. The effect of different dosing regimens of motesanib on the gallbladder: a randomized phase 1b study in patients with advanced solid tumors. BMC Cancer. 2013 May 16;13:242. doi: 10.1186/1471-2407-13-242. PMID 23679351
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com